CLINICAL TRIAL: NCT02091583
Title: Developing and Evaluating a Novel Food Supplement, Consisting of Canola Oil, Fibre and DHA, Aiming at the Management of CVD Risk in a Population With Metabolic Syndrome
Brief Title: Canola Oil, Fibre and DHA Enhanced Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Agriculture and Agri-Food Canada (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: B2014:029
Record Dates: First submitted 2014-03-12; First posted 2014-03-19 (Estimated); Last update posted 2023-03-17 (Actual); Status verified 2021-04

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome; Cardiovascular disease; High Oleic Canola Oil; DHA; β-glucan; Barley; Cholesterol; Lipoproteins; Lipids; Inflammation; Glucose; Insulin; Satiety; Body composition; Blood pressure
MeSH Terms: conditions — Metabolic Syndrome; Cardiovascular Diseases; Inflammation; Insulin Resistance | interventions — Butter; Safflower Oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Butter, sunflower and safflower oil (Placebo Comparator): The oil (50g/day) is given in muffin and cookies made with refined wheat flour (3 g/day)daily for 4 weeks.
  Interventions: Dietary Supplement: Butter, sunflower and safflower oil
- High Oleic Canola Oil and DHA (HOCO-DHA) (Active Comparator): The oil (50g/day) is given in muffin and cookies made with refined wheat flour (3 g/day) daily for 4 weeks.
  Interventions: Dietary Supplement: High Oleic Canola Oil and DHA (HOCO-DHA)
- Barley Beta-glucan (Active Comparator): The Barley beta-glucan (3 g/day) is given in muffin and cookies made with a combination of butter, sunflower and safflower oil (50 g/day) daily for 4 weeks.
  Interventions: Dietary Supplement: Barley beta-glucan
- HOCO-DHA and Barley beta-glucan (Active Comparator): The oil and beta-glucan (50g and 3g/day, respectively) is given in muffin and cookies daily for 4 weeks.
  Interventions: Dietary Supplement: HOCO-DHA and Barley beta-glucan

INTERVENTIONS:
Dietary Supplement: Butter, sunflower and safflower oil
  Arms: Butter, sunflower and safflower oil
Dietary Supplement: High Oleic Canola Oil and DHA (HOCO-DHA)
  Arms: High Oleic Canola Oil and DHA (HOCO-DHA)
Dietary Supplement: Barley beta-glucan
  Arms: Barley Beta-glucan
Dietary Supplement: HOCO-DHA and Barley beta-glucan
  Arms: HOCO-DHA and Barley beta-glucan

SUMMARY:
The purpose of this study is to examine the effects of consumption of a novel food supplement consisting of Canola Oil, Fibre and DHA, containing the most effective food bioactives, including n-3 fatty acid enriched dietary oil high in monounsaturated fatty acids (MUFAs) and soluble dietary fibre, aiming at the management of heart disease risk factors in people with metabolic syndrome and to test its efficacy and safety in humans.

DETAILED DESCRIPTION:
The proposed study is a randomized, single-blind, crossover trial, it will be conducted at the Richardson Centre for Functional Food and Nutraceuticals (RCFFN), University of Manitoba. The study design will consist of 4 phases with 30 days per phase, each phase will be separated by 4-week washout periods. Participants will consume a recommended weight-maintaining diet (35% energy from fat, 50% carbohydrate, 15% protein) supplemented with the following novel Muffin and cookies: (a) control food containing butter, sunflower and safflower oil comprised largely of saturated fat with substantial levels of n-6 linoleic acid, and refined wheat flour common to current North American intakes, (b) food containing high oleic canola oil and docosahexaenoic acid (HOCO-DHA) and refined wheat flour, (c) food containing high molecular weight barley B-glucan and a combination of sunflower, safflower oil and butter, (d) food containing combination of HOCO-DHA and high molecular weight barley β-glucan. Treatments will be isocalorically incorporated into muffin and cookies consumed in equal parts at breakfast and supper.

ELIGIBILITY:
Inclusion Criteria:

* BMI≥25 Kg/m2
* Waist circumference ≥94 cm (males) or ≥80 cm (females)

Meet at least two of the following:

* Triglycerides ≥1.7 mmol/L
* High density lipoprotein (HDL) cholesterol <1 mmol/L (males) or <1.3 mmol/L (females)
* Low density lipoprotein (LDL) cholesterol ≥2.7 mmol/L
* Fasting glucose ≥5.6 mmol/L

Exclusion Criteria:

* Consuming lipid lowering medications
* Consuming nutritional supplements
* Disease or disorder that could interfere with absorption
* Smokers
* Hypertension ≥150 mmHg (systolic) and/or ≥100 mmHg (diastolic)
* Planning to become pregnant
* Consume >1 alcoholic drink/day
* Medication within a month prior to screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Change in 10-year Framingham CVD risk score | The 10-year Framingham CVD risk score will be calculated for each participant at the end of each four 4-week treatment phases over a period of seven months
  Change in 10-year Framingham CVD risk will be assessed using the multivariable Framingham risk equation.

SECONDARY OUTCOMES:
Change in blood lipid profile (TC, TG, LDL-C, HDL-C) | Blood samples will be collected at the start and end of each of the four 4-week treatment phases over a period of seven months
  Lipid profile will be determined using the automated enzymatic methods. Subfractions and particle size of LDL-C and HDL-C will be determined by LipoprintR system.
Change in inflammatory markers | Blood samples will be collected at the start and end of each of the four 4-week treatment phases over a period of seven months
  Determination of inflammatory markers and cytokines will be measured by commercially available ELISA kits.
Cholesterol synthesis rate | Fasting blood samples will be collected during the last 2 days of the four 4-week treatment phases over a period of seven months
  Participants will be asked to consume deuterium oxide (D2O) at the end of each phase. In addition, on day 29 a fasting baseline blood sample is taken prior to administration of an oral dose of D2O as tracer to measure fractional cholesterol synthesis. Fasting blood samples will be obtained 24 h following the tracer dose on day 30.
Change in body composition | Measurements will be done at the beginning and end of each of the four 4-week treatment phases over a period of seven months
  Changes in body composition will be assessed using dual-energy X-ray absorptiometry (DXA) scans. In addition, body weight, waist and hip circumferences will be measured.
Blood Pressure | Measurements will be done at the beginning and end of each of the four 4-week treatment phases over a period of seven months
  Blood pressure data (change in both systolic and diastolic) was taken 4 times at 2-minutes intervals. The last 3 measurements will be averaged.
Fasting plasma insulin concentration | Blood samples will be collected at the start and end of each of the four 4-week treatment phases over a period of seven months
  Insulin homeostasis modelling assessment will be utilised as an estimate for % β-cell function and insulin resistance.
Plasma and RBC fatty acid analysis | Blood samples will be collected at the start and end of each of the four 4-week treatment phases over a period of seven months
  Plasma and RBC total lipids will be extracted using the Folch method involving chloroform-methanol (2:1, v/v) containing 0·01% BHT and heptadecanoic acid as an internal standard. Extracted fatty acids will be methylated with methanolic HCl. Fatty acid methyl esters will be separated on a Supelcowax 10 column using a gas chromatograph equipped with a flame ionisation detector .
Microbiome analysis | Fecal samples will be collected at the start and end of each of the four 4-week treatment phases over a period of seven months
  Bacterial DNA from the fecal samples will be extracted using ZR Fecal DNA MiniPrepTM kit and DNA concentration along with quality will be determined using a NanoDrop 2000c.The gut microbial composition will be analysed by next generation Illumina based sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Peter JH Jones, PhD, Study Chair — Richardson Centre for Functional Foods and Nutraceuticals, University of Manitoba; Nancy Ames, PhD, Principal Investigator — Agriculture and Agri-Food Canada; Vanu R Ramprasath, PhD, Principal Investigator — Richardson Centre for Functional Foods and Nutraceuticals, University of Manitoba; Sijo Joseph, PhD, Principal Investigator — Agriculture and Agri-Food Canada
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Ramprasath VR, Thandapilly SJ, Yang S, Abraham A, Jones PJ, Ames N. Effect of consuming novel foods consisting high oleic canola oil, barley beta-glucan, and DHA on cardiovascular disease risk in humans: the CONFIDENCE (Canola Oil and Fibre with DHA Enhanced) study - protocol for a randomized controlled trial. Trials. 2015 Oct 31;16:489. doi: 10.1186/s13063-015-1014-5. PMID 26518870